CLINICAL TRIAL: NCT06718634
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-M08D1 for Injection in Patients With Relapsed or Refractory Lymphoid Malignancies
Brief Title: A Study of BL-M08D1 in Patients With Relapsed or Refractory Lymphoid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M08D1-102
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Lymphoid Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M08D1 (Experimental): Participants receive BL-M08D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M08D1

INTERVENTIONS:
Drug: BL-M08D1 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter, dose-escalation and extended-enrollment, nonrandomized phase I study to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of BL-M08D1 for injection in relapsed or refractory lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Recurrent or refractory lymphoid malignancies confirmed by histopathology and/or cytology that are incurable or for which no standard treatment is currently available;
6. Consent to provide archival tumor tissue samples or fresh tissue samples from primary or metastatic lesions within 2 years;
7. ECOG≤2;
8. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
10. Organ function level must meet the requirements;
11. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
12. Urinary protein ≤2+ or ≤1000mg/24h;
13. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients (regardless of male or female) should use adequate barrier contraception during the whole treatment cycle and for 6 months after the end of treatment;
14. Subjects were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Chemotherapy, biological therapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Palliative radiotherapy or traditional Chinese medicine with anti-tumor indications within 2 weeks before the first dose;
2. History of severe heart disease;
3. QT prolongation, complete left bundle branch block, III degree atrioventricular block;
4. Active autoimmune and inflammatory diseases;
5. Other malignant tumors diagnosed within 5 years before the first dose;
6. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
7. Patients with poor glycemic control or with diabetic gangrene;
8. A history of ILD requiring steroid therapy or current ILD or grade ≥2 radiation pneumonitis;
9. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
10. Patients with central nervous system involvement;
11. Had a history of or central nervous system disease;
12. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any component of BL-M08D1 excipients;
13. Received previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
14. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
15. Active infection requiring systemic therapy within 4 weeks before the first dose of study drug;
16. Pleural, abdominal, pelvic or pericardial effusion requiring drainage and/or with symptoms within 4 weeks before the first dose of study drug;
17. Received another trial drug 4 weeks or 5 half-lives before the first dose;
18. Pregnant or lactating women;
19. Other conditions for participation in the trial were not considered appropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M08D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M08D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M08D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M08D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M08D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M08D1 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-M08D1 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M08D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M08D1 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China